CLINICAL TRIAL: NCT05087849
Title: Therapeutic Intralesional Nonavalent HPV Vaccine for Genital Condylomata in Adults: an Open Label Pilot Study
Brief Title: Intralesional HPV Vaccine for Condylomata
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-35086
Record Dates: First submitted 2021-10-08; First posted 2021-10-21 (Actual); Results first posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Human Papilloma Virus; Warts; Warts, Genital; Condyloma; Condylomata Acuminata
Keywords: Gardasil 9; nonavalent human papillomavirus vaccine; intralesional immunotherapy; condyloma; genital warts
MeSH Terms: conditions — Warts; Condylomata Acuminata | interventions — Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Intervention Model Description: This is an open-label, single-arm study in which all participants will receive intralesional Gardasil 9 vaccine to their condyloma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intralesional injection of nonavalent human papillomavirus vaccine (Experimental): Single-arm, open-label study. Intervention consists of intralesional injection of nonavalent human papillomavirus vaccine at 0 and 4 weeks.
  Interventions: Biological: nonavalent human papillomavirus vaccine

INTERVENTIONS:
Biological: nonavalent human papillomavirus vaccine — Intralesional injection of nonavalent human papillomavirus vaccine (Gardasil 9) at 0 and 4 weeks

SUMMARY:
This study will investigate whether injecting genital warts with small quantities of the Gardasil 9 vaccine has an effect on the warts.

DETAILED DESCRIPTION:
This is a prospective, open-label, proof-of-concept research study to assess the effectiveness of intralesional nonavalent in the treatment of patients with genital condylomata. The study will be conducted at Zuckerberg San Francisco General Hospital. The planned intervention is to provide 10 subjects with at least 3 genital condylomata with intralesional nonavalent human papillomavirus vaccine (Gardasil 9) at 0 and 4 weeks. Then, the study subjects will be followed for a further 8 weeks to monitor for change in wart size and wart number.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all genders aged ≥ 18 years
* Signed informed consent form
* Confirmed clinical diagnosis of genital condylomata with minimum of 3 genital condylomata, each measuring >3mm
* Individuals who are able to become pregnant will be advised on the following:

All individuals who are able to become pregnant will be asked about their reproductive health, sexual activity (partners, practices, prevention of pregnancy) and be advised that administration of vaccine during pregnancy is not recommended while data collection to monitor pregnancy and infant outcomes following exposure to the papillomavirus (9-valent) vaccine is ongoing. However, based on available data, an increased risk of adverse pregnancy outcomes, specifically miscarriage or congenital anomalies, has not been observed following inadvertent administration of the papillomavirus vaccine during pregnancy. Individuals who are able to become pregnant are advised to contact us immediately and will not receive any further intralesional vaccine.

Exclusion Criteria:

* Participants will be asked about pregnancy at time of recruitments. Individuals who are pregnant or are planning to become pregnant will not be permitted to participate in the study, as ACOG does not recommend Gardasil 9 during pregnancy. Participants will be encouraged not to participate in the study if they believe they may become pregnant during the study.
* Participants will be asked about allergic reaction to yeast and vaccine components at time of recruitment. Subjects with severe allergic reactions to baker's yeast (Saccharomyces cerevisiae, a vaccine component), or other vaccine components (ie polysorbate 80, Merck amorphous aluminum hydroxyphosphate sulfate) will not be permitted to participate in this study.
* Participants' vaccination history will be reviewed at time of recruitment. Patients who have previously received any prior human papillomavirus vaccine will not be permitted to participate in this study.
* Subjects' medical history and current medications will be reviewed at time of recruitment. Subjects taking immune suppressive medications (steroids such as prednisone or dexamethasone, immunosuppressive agents such as methotrexate, azathioprine, cyclosporine, immunomodulatory agents such as apremilast, or immunomodulatory biologic agents such as adalimumab, guselkumab or ustekinumab) will be excluded. Subjects with medical conditions that significantly alter the immune system, such as known HIV infection, leukemia or lymphoma will be excluded from this pilot study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayan Kusari, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intralesional Injection of Nonavalent Human Papillomavirus Vaccine
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intralesional Injection of Nonavalent Human Papillomavirus Vaccine
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants] — Age
  Participants
    <=18 years | 0
    Between 18 and 65 years | 2
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Wart Number
Description: Change in number of warts in genital area.
Time Frame: Baseline (week 0) and Week 12.
Measure: Mean (Standard Deviation); unit: warts
Groups:
- All Subjects: Single-arm.
Arm/Group | All Subjects
Number analyzed (Participants) | 2
warts | 0.5 (0.5)

2. Primary Outcome: Change in Average Size of Genital Warts in mm
Description: Mean size of warts in genital area, as measured by study personnel at study visits .
Time Frame: to be measured at baseline (week 0) and Week 12
Measure: Mean (Standard Deviation); unit: mm
Groups:
- All Subjects: All subjects in study
Arm/Group | All Subjects
Number analyzed (Participants) | 2
mm | 0.13 (0.65)

3. Secondary Outcome: Change in Score of Specific Questionnaire for Condylomata Acuminata (CECA)
Description: Established tool to measure quality of life with respect to condyloma. Will be administered at baseline and week 12 by study personnel. It comprises 10 items and 2 dimensions. The emotional dimension includes 6 items and the sexual activity dimension includes 4 items. The questions refer to the past 7 days. The higher the score the better the quality of life. The global scoring range was 10-50, ranging from 6 to 30 in the emotional dimensions and from 4 to 20 in the sexual activity dimension.
Time Frame: to be measured at baseline (week 0) and week 12
Population: All subjects
Measure: Mean (Standard Deviation); unit: CECA score
Arm/Group | All Subjects
Number analyzed (Participants) | 2
CECA score | -18.5 (1.5)

4. Secondary Outcome: Change in Score of Dermatology Quality of Life Index (DLQI)
Description: Established tool to measure quality of life with any dermatologic disease. Will be administered at baseline and week 12 by study personnel. Consists of 10 questions scored from 0-3. The DLQI is calculated by adding the score of each question, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Time Frame: to be measured at baseline (week 0) and week 12
Measure: Mean (Standard Deviation); unit: DLQI score
Arm/Group | All Subjects
Number analyzed (Participants) | 2
DLQI score | 0 (2)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intralesional Injection of Nonavalent Human Papillomavirus Vaccine
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-03-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT05087849/Prot_SAP_ICF_001.pdf